CLINICAL TRIAL: NCT03802838
Title: Clinical Evaluation of Acupuncture Treatment for Negative Symptoms of Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZHYY-ZXYJHZX-2-201708
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2018-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia ，acupuncture，Amisulpride
MeSH Terms: conditions — Schizophrenia | interventions — Acupuncture Therapy; Amisulpride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Active Comparator): Acupuncture+Amisulpride
  Interventions: Device: acupuncture; Drug: Amisulpride
- Amisulpride (Other): Amisulpride only.
  Interventions: Drug: Amisulpride

INTERVENTIONS:
Device: acupuncture — Schizophrenia with negative symptoms were treated with Amisulpride, and the patients still remained negative symptoms and cognitive impairment.Amisulpride is allowed in a dose range of 50-1200 mg / d, once or twice a day for at least 12 weeks. These patients were combined with acupuncture. Acupuncture points include:'Yintang', 'Shenting', 'Taiyang', 'Jingming', 'Zanzhu', 'Yuyao', 'Jiaosun', 'Baihui', 'Fengchi', 'Anmian'.
  Arms: Acupuncture
Drug: Amisulpride — Schizophrenia with negative symptoms were treated with Amisulpride, and the patients still remained negative symptoms and cognitive impairment.Amisulpride is allowed in a dose range of 50-1200 mg / d, once or twice a day for at least 12 weeks.

SUMMARY:
To explore the effects of combined traditional Chinese and Western medicine( Chinese acupuncture combined with Amisulpride Tablets) on negative symptoms, cognitive function and social function in patients with schizophrenia, and the side effects and safety of Chinese acupuncture combined with Amisulpride Tablets.

DETAILED DESCRIPTION:
Our research hypothesis：1. Medically assisted Acupuncture in schizophrenia can improve negative symptoms；2. Drug assisted Acupuncture Therapy has better cognitive function in schizophrenic patients than single drug；3. Schizophrene with acupuncture have fewer and lighter adverse reactions。This study was carried out only in Shanghai Mental Health Center. It was a parallel randomized study.Schizophrene with negative symptoms were treated with atypical antipsychotic drug amisulpride, but still remained negative symptoms. Using the mature Chinese medicine therapy acupuncture auxiliary treatment, using the more reliable clinical evaluation method (the grader blind method: The raters were not sure which patients were the study group or the control group), compared with the single drug treatment, To observe the changes of negative symptoms and cognitive function, and the incidence of adverse reactions of acupuncture therapy, to explore the "new" auxiliary means for the treatment of negative symptoms, to guide clinical individualization and accurate medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of schizophrenia according to International classification diagnosis-10(ICD-10)
* patients at an age between 18～60 years old of Han nationality

Exclusion Criteria:

* other psychiatric diagnoses
* Suffering from serious physical disease and can not accept the treatment
* Patients to be diagnosed according to ICD-10 for substance abused, development delayed
* Inability to sign informed consent because of capacity due due to severe mental illness, significant psychomotor agitation or slowness test completion
* claustrophobic
* metal implantation in vivo

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
The Positive and Negative Syndrome Scale (PANSS) | the baseline
  a 30-items, 7-point rating scale; the 7 rating points represent increasing levels of psychopathology: 1= absent, 2= minimal, 3= mild, 4 = moderate, 5= moderate-severe, 6= severe, 7= extreme; of the 16 items, 7 were chosen to constitute Positive Scale, 7 items for Negative Scale and the remaining 16 items for a General Psychopathology Scale
The Positive and Negative Syndrome Scale (PANSS) | the end of 12 weeks
  a 30-items, 7-point rating scale; the 7 rating points represent increasing levels of psychopathology: 1= absent, 2= minimal, 3= mild, 4 = moderate, 5= moderate-severe, 6= severe, 7= extreme; of the 16 items, 7 were chosen to constitute Positive Scale, 7 items for Negative Scale and the remaining 16 items for a General Psychopathology Scale
The Clinical Assessment Interview for Negative Symptoms (CAINS) | the baseline
  including CAINS and CAINS self-reported checklists
The Clinical Assessment Interview for Negative Symptoms (CAINS) | the end of 12 weeks
  including CAINS self-reported checklists
Repeatable sets of neuropsychological state measurements (RBANS) | the baseline
  That allows us to measure cognitive impairment in patients.
Repeatable sets of neuropsychological state measurements (RBANS) | the end of 12 weeks
  That allows us to measure cognitive impairment in patients.

SECONDARY OUTCOMES:
The Temporal Experience of Pleasure Scale (TEPS) | the baseline
  That allows us to measure the experience of pleasure in patients.
The Temporal Experience of Pleasure Scale (TEPS) | the end of 12 weeks
  That allows us to measure the change of experience of pleasure in patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenghui YI, Principal Investigator — SHANGHAI MENTAL HEALTH CENTRE
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No